CLINICAL TRIAL: NCT01404260
Title: Intercalating and Maintenance Use of Iressa vs. Chemotherapy in Selected Advanced NSCLC: a Randomised Study
Brief Title: Intercalating and Maintenance Use of Iressa Versus Chemotherapy in Selected Advanced Non Small Cell Lung Cancer
Acronym: ISCAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: The First Hospital of Jilin University (Other); Ruijin Hospital (Other); Fudan University (Other); Jiangsu Cancer Institute & Hospital (Other); Nanjing PLA General Hospital (Other); Wuxi No. 4 People's Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Henan Cancer Hospital (Other Government); Changhai Hospital (Other); NanJing PLA 81 Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Lu shun, Director of Department Shanghai Lung Tumor Clinical Center, Shanghai Chest Hospital, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG 1102
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: chemotherapy; maintenance therapy; gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine +Carboplatin +Gefitinib (Experimental): Arm A: Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum 4 cycles, Gefitinib 250mg/d every cycle d15-25, and Gefitinib 250mg/d from d15 of last cycle until disease progression
  Interventions: Drug: Gefitinib; Drug: Gemcitabine +Carboplatin
- Gemcitabine +Carboplatin (Active Comparator): Arm B: Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum4 cycles, observation until disease progression
  Interventions: Drug: Gemcitabine +Carboplatin

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg/d every cycle d15-25,and Gefitinib 250mg/d from d15 of last cycle until disease progression
  Other Names: Iressa
  Arms: Gemcitabine +Carboplatin +Gefitinib
Drug: Gemcitabine +Carboplatin — Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum 4 cycles

SUMMARY:
Platinum-based combination chemotherapy, such as gemcitabine-carboplatin, is one of the standard first-line therapy for advanced non-small cell lung cancer (NSCLC).

Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI) have clinical efficacy, as compared with the best supportive care or standard chemotherapy, when given as second-line or third-line therapy for advanced NSCLC.

Treatment with EGFR-TKI is most effective in female, never-smoker, or patients with adenocarcinoma, and patients of Asian origin. In these populations, such treatment is associated with favorable objective response rates, progression-free survival, and overall survival. These populations also have a relatively high incidence of somatic mutations in the region of the EGFR gene that encodes the tyrosine kinase domain.

The recent study(IPASS) by Tony S. Mok showed gefitinib was superior to carboplatin-paclitaxel as an initial treatment for pulmonary adenocarcinoma among nonsmokers or former light smokers in East Asia . In the subgroup of 261 patients who were positive for the EGFR gene mutation, PFS was significantly longer among those who received gefitinib than among those who received carboplatin-paclitaxel(HR= 0.48,P<0.001), whereas in the subgroup of 176 patients who were negative for the mutation, PFS was significantly longer among those who received carboplatin-paclitaxel(HR=2.85,P<0.001). Gefitinib treatment was well tolerated, with lower in hematologic toxicity, and no treatment-related interstitial lung disease.In this study(IPASS), only patients with a mutation of the EGFR gene in the tumor could get benefit from gefitinib as first line treatment.

Tony S. Mok and his colleague also found that intercalating and maintenance administration of erlotinib(another EGFR-TKI)following gemcitabine/platinum chemotherapy as first line therapy led to a significant improvement in PFS .

DETAILED DESCRIPTION:
Nowadays,EGFR mutation status is unknown for most of the advanced NSCLC patients in clinical practice.Those patients with high probability of EGFR mutation maybe could get benefit from gefitinib as first-line treatment. For this reason, the investigators need more investigation to focus on EGFR mutation unknown patients. In the previous study (including FAST-ACT), the patients enrolled trial received EGFR-TKI plus chemotherapy nearly simultaneously,so the investigators could not know whether those patients gained benefit from EGFR-TKI or chemotherapy, maybe chemotherapy alone was enough. If the patients with EGFR mutation status unknown could get stable disease(SD) after two cycles of chemotherapy,those patients may be optimal for the investigation of intercalating and maintenance administration of gefitinib. The reasons are that chemotherapy may be enough for those with objective response after two cycles chemotherapy, of course, those with disease progression (PD) should be excluded from the study.

On the basis of these and other studies, the investigators hypothesized that in a selected population,first-line chemotherapy(gemcitabine +carboplatin) with intercalating and maintenance use of gefitinib would be more efficacious than chemotherapy alone. In this study, the investigators compared the efficacy, safety, and adverse-event profile of chemotherapy plus gefitinib with those of chemotherapy alone, when these drugs were used as first-line treatment in nonsmokers or former light smokers in China, who had lung adenocarcinoma with EGFR gene mutation unknown.

ELIGIBILITY:
Inclusion Criteria:

* After two cycles chemotherapy(gemcitabine plus carboplatin), patients with stable disease(SD) by RECIST1.1.
* Patients between 18 and 75 years of age.
* Present with histologically proven or cytological diagnosis of adenocarcinoma NSCLC Stage IIIB or IV as defined by the American Joint Committee on Cancer Staging Criteria for Lung Cancer, that is not amenable to curative therapy,such as surgery or radiotherapy and so on.
* No prior systemic chemotherapy or targeted therapy for lung cancer before screening.
* Never smokers(defined as having smoked less than 100 cigarettes in their lifetime ) or light ex-smokers (defined as having ceased smoking at least 15 years before Day 1 of study treatment and having smoked 10 pack-years or fewer).
* EGFR mutation status unknown.
* ECOG performance status of 0 or 1.
* Adequate organ function.
* Prior radiation therapy allowed to <25% of the bone marrow . Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study enrollment. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment.
* Signed informed consent document on file.
* Estimated life expectancy of ≥12 weeks.
* Patient compliance and geographic proximity that allow adequate follow up.

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib.
* Sympotomatic patients with brain metastases.
* Pleural effusion or pericardiac effusion that cannot be controlled by drainage or other procedures.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Interstitial pneumonia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD., Principal Investigator — Guangdong Province Clinical Trial Association
Locations (1):
- Shanghai Lung Tumor Clinical Center,Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Gefitinib + Gemcitabine + Carboplatin: Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum 4 cycles, Gefitinib 250mg/d every cycle d15-25, and Gefitinib 250mg/d from d15 of last cycle until disease progression
- Arm B: Gemcitabine + Carboplatin: Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum4 cycles, observation until disease progression
Period: Overall Study
Arm/Group | Arm A: Gefitinib + Gemcitabine + Carboplatin | Arm B: Gemcitabine + Carboplatin
Started | 109 | 110
Completed | 106 | 101
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Arm A: gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum 4 cycles, gefitinib 250mg/d every cycle d15-25, and gefitinib 250mg/d from d15 of last cycle until disease progression
  gefitinib: gefitinib 250mg/d every cycle d15-25,and gefitinib 250mg/d from d15 of last cycle until disease progression
- Arm B: gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum4 cycles, observation until disease progression
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 109 | 110 | 219
Age, Continuous [Median (Full Range); unit: Years] | 56 [49 to 62] | 58 [50 to 63] | 57 [49 to 63]
Gender [Count of Participants; unit: Participants]
  Female | 88 | 83 | 171
  Male | 21 | 27 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 109 | 110 | 219
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 109 | 110 | 219

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or progression in existing non-target lesions,or the appearance of one or more new lesions .
Time Frame: The evaluation of disease is demanded every two months for the patients receiving maintenance use of Gefitinib or patients in observation after chemotherapy,until disease progression occured
Population: Efficacy analysis, including PFS will be based on intent to treat (ITT) population.. ITT population includes all the randomised patients who receive at least one dose of study treatment with at least one baseline data of volume of plaque and at least one data after treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A: Gefitinib+Gemcitabine +Carboplatin: Arm A: Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum 4 cycles, Gefitinib 250mg/d every cycle d15-25, and Gefitinib 250mg/d from d15 of last cycle until disease progression
- Arm B: Gemcitabine +Carboplatin: Gemcitabine 1250mg/m2+Carboplatin AUC=5, every 4 weeks, maximum4 cycles, observation until disease progression
Arm/Group | Arm A: Gefitinib+Gemcitabine +Carboplatin | Arm B: Gemcitabine +Carboplatin
Number analyzed (Participants) | 106 | 101
months | 9.7 [5.9 to 11.3] | 4.2 [3.6 to 4.7]

ADVERSE EVENTS:
Time Frame: 4years
Description: Safety analysis included all patients who received at least one dose of the study drug and had at least one follow-up safety assessment. Safety assessments were analyzed mainly using descriptive statistics.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 14/109 | 5/110
Other Adverse Events (participants affected / at risk) | 9/109 | 1/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=109) | Arm B (N=110)
Leukopenia (Blood and lymphatic system disorders) | 14 (17) | 5 (26)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=109) | Arm B (N=110)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less